CLINICAL TRIAL: NCT02576041
Title: Effects of Bilastine on F1 Simulator Driving Performance in Patients Affected by Allergic Rhinitis and/or Urticaria
Acronym: F1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEIN/14/Bil-ARU/001; 2015-001313-26 (EudraCT Number)
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Allergic Rhinitis; Urticaria
Keywords: driving simulator
MeSH Terms: conditions — Rhinitis, Allergic; Urticaria | interventions — bilastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (run-in); Bilastine (Experimental): At V0, the enrolled patient received the complete drug-kit and started a 7 (+3)-day wash-out period with placebo. At the end of the 7 (+3)-days of placebo-treatment period, patients repeated the F1-high speed simulator test at Visit V1, and afterwards initiated the 7 (+3)-day treatment period with active treatment (bilastine).
  Interventions: Drug: Bilastine; Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — Bilastine tablets once a day for 7+3 days
  Other Names: Robilas
Drug: Placebo — Placebo tablets once a day during 7+3 days run in period

SUMMARY:
The aim of the study is to evaluate the effects of Bilastine on patients' attention and reactivity levels by measuring psychophysical performance at a F1-high speed simulator driving test.

DETAILED DESCRIPTION:
This was a phase IV, interventional, prospective, mono-centric, single arm, uncontrolled, open label trial. The study included outpatient affected by Allergic Rhinitis and/or Chronic Urticaria, responding to inclusive criteria and able to perform a preliminary driving test on F1-high speed simulator (at the simulator centre) without experiencing signs or symptoms of intolerance towards the drive simulation (e.g., nausea, vomiting or dizziness etc). Each subject underwent 3 ambulatory visits at the hospital site and 3 driving test at the simulator centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by allergic rhinitis (seasonal or perennial) or urticaria (induced and not induced) who need histamine H1-receptor antagonist therapy according to PI therapeutic decision;
* Males and females aged between 21 and 55 years;
* Body Mass Index (BMI) between 19 and 30 kg/m2 (included);
* If women: negative pregnant test and contraception from at least 30 days before the study (Visit V-1) and up to the end of the study. For women patients the negative pregnant test will be acquired before the Simulator performance (Visit V-1H);
* Subjects having a valid driving license from more than 3 years;
* Subjects having a driving experience of at least 5000 km per year;
* Subjects able to understand the protocol and to come to the visits;
* Subjects able to give a written informed consent;
* Subjects who, at investigator's judgment, are likely to be compliant during the study and do not use potentially adulterating drugs;
* Potential compliant subjects will be enrolled only if they tolerate driving the F1-simulator (starting from V-1 S).

Exclusion Criteria:

* Subjects with autoimmune urticaria;
* Hypersensitivity to the active substance bilastine or to any of the excipients;
* History or symptoms of severe mental or physical disorders or taking substance and alcohol;
* Excessive smoking (more than 20 cigarettes per day), or consumption of caffeinated beverages (more than 6 cups per day);
* Subjects who need unimpaired psychophysical condition due to their job;
* Subjects with any non corrected visual defect or locomotor disorder which could interfere with the study;
* Subjects ineligible at Visit V-1;
* Subjects with known allergic reactions to antihistamines;
* Subjects with porphyria;
* Subjects with important sleep disturbances or kinetosis;
* Subjects with clinically important (based on Investigator's judgment) renal or hepatic impairment, or gastrointestinal diseases (e.g. malabsorption);
* Subjects with a medical history of seizure (i.e. epileptic related) or with current seizure;
* Presence of significant medical condition/concomitant illnesses that, in the opinion of the Investigator, renders the patient immunocompromised or not suitable for a clinical trial or could adversely affect the subject's participation or evaluation in this study;
* Subjects for whom, in the opinion of the Investigator, there is concern about compliance with the study procedures;
* Presence of a permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhoea diseases, congenital malformations or surgical mutilations of the gastrointestinal tract);
* Presence of active cancer which requires chemotherapy or radiation therapy;
* Presence of alcohol abuse or drug addiction;
* Pregnancy or breast-feeding;
* Treatment with: diuretics, corticosteroids (other than medication applied topically), central nervous system medications or medications with sedative effects (sleep inducing or antidepressant, sedative medications), medications that can interact with bilastine, other medications. In particular, patients treated with any of the following drugs will be excluded:

  * Imipramine antidepressants, anticholinergic antiparkinsonians, atropine antispasmodics, disopyramide, phenothiazine neuroleptics;
  * Sedative antidepressants, monoamine oxidase (MAOI) inhibitors, barbiturates, benzodiazepines, clonidine and related substances, hypnotics, morphine derivatives (analgesics, antitussives, replacement treatments), neuroleptics, anxiolytics;
  * Treatments with P-glycoprotein inhibitors (e.g. ketoconazole, erythromycin, cyclosporine, ritonavir, diltiazem), which may increase the plasmatic levels of bilastine;
  * Treatments that are substrates or inhibitors of OATP1A2 (e.g. ritonavir, rifampicin), which may decrease plasma concentrations of bilastine
  * Other treatments that can interact with bilastine (e.g. ketoconazole, erythromycin, diltiazem); Treatment with anticoagulants (e.g. warfarin);
  * Sedatives, hypnotics, tranquillizers or any other addictive agents;
  * Other treatments not admitted during the study: betahistine, anticholinesterases, arrhythmogenic drugs;
  * H2-antihistamines;
  * H1 antihistamines other than study medication or rescue medication. In any case, the possibility of inclusion of patients taking any of these drugs will be left at the Investigator's judgment.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Pepe, Principal Investigator — Allergology Unit, Azienda Ospedaliero-Universitaria Policlinico di Modena
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening was performed in 2 separate sections, at hospital site (H) and at the simulator (S) center. A total of 19 patients were screened and only one discontinued study before starting placebo treatment due to agitation, sickness, transpiration and vomiting at the simulator driving test.
Period: Placebo (run-in)
Arm/Group | Placebo (run-in); Bilastine
Started | 18
Completed | 18
Not Completed | 0
Period: Bilastine (Active Treatement)
Arm/Group | Placebo (run-in); Bilastine
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Placebo (run-in); Bilastine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 18

OUTCOME MEASURES:

1. Primary Outcome: Standard Deviation Lateral Position (SDLP) Evaluated During the F1 Simulator Test
Description: SDLP (mainly assessing attention capacities). This is a measure of weaving and quality in keeping the requested path. The vehicle position was constantly monitored. The deviation from central position was registered.
Time Frame: 7+3 days of active treatment
Population: The study included adult outpatient of either sex affected by allergic rhinitis (seasonal or perennial) and/or chronic urticaria (induced or not induced) able to perform a preliminary driving test on F1-high speed simulator without experiencing sign or symptoms of intolerance towards the drive simulation (e.g. nausea, vomiting or dizziness).
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Bilastine: Patients repeated the F1-high speed simulator test at Visit V1, and afterwards initiated the 7 (+3) day treatment period with Bilastine
Arm/Group | Bilastine
Number analyzed (Participants) | 18
meters | -0.041 (0.047)

2. Secondary Outcome: Maintenance of Constant Speed Evaluated During the F1 Simulator
Description: Different speed were maintained as requested by the simulator. Variations during the test were recorded. The mean deviation from the requested speed was registered.
Time Frame: 7±3 days of active treatment
Population: The study included adult outpatient of either sex,affected by Allergic Rhinitis (seasonal or perennial) and/or Chronic Urticaria (induced or not induced),able to perform a preliminary driving test on F1-high speed simulator without experiencing signs or symptoms of intolerance towards the drive simulation (e.g. nausea, vomiting or dizziness, etc).
Measure: Mean (Standard Deviation); unit: Km/h
Arm/Group | Bilastine
Number analyzed (Participants) | 18
Km/h | -1.397 (2.991)

3. Secondary Outcome: Time to Reaction Evaluated During the F1 Simulator
Description: During the test, at different times, the patient will be requested (by led enlighten on the dashboard) to execute actions on the steering-wheel. The delay in executing the requested actions will be registered.
Time Frame: 7±3 days of active treatment
Population: Adult outpatient of eighter sex affected by Allergic Rhinitis (seasonal or perennial) and/or chronic urticaria (induced or not induced) able to perform a preliminary driving test on F1-high speed simulator without experiencing sign or symptoms of intolerance towards the drive simulation (e.g. nausea, vomiting or dizziness).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Bilastine
Number analyzed (Participants) | 18
msec
  Time reaction to Button A | -34.5 (95.71)
  Time reaction to button B | -18.25 (66.28)

ADVERSE EVENTS:
Arm/Group | Placebo (run-in); Bilastine
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (run-in); Bilastine (N=18)
bradycardia (Cardiac disorders) | 1 (1)
Laboratory test abnormal (Investigations) | 17 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can disclose the results after sending to the Sponsor, for appropriate knowledge and / or possible review, copy of the document, at least 90 days prior to publication and / or presentation. If requested in writing by the Sponsor, the PI will agree to make changes to the manuscript and / or deferred publication of the manuscript further 90 days to allow the patent application.